CLINICAL TRIAL: NCT01183052
Title: Mitochondrial Respiratory Chain and Peripheral Muscle Dysfunction in COPD Patients
Brief Title: Mitochondrial Dysfunction and Oxidative Stress in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Santé (Other)
Collaborators: Centre Hospitalier Régional Universitaire Montpellier (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2009-A00426-51
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: COPD Patients
Keywords: COPD; exercise tolerance; oxidative stress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training (Other): 20 sessions of training
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — 20 sessions of training
  Other Names: CT

SUMMARY:
The purpose of this study is to understand the underlying mechanisms of improved exercise tolerance in COPD patients after training program.

DETAILED DESCRIPTION:
Training protocol used is based on recommendations (Nici et al., 2006) and was previously used in our group (Varray et al., 1991; Vallet et al., 1997). A minimum of 20 sessions in 4-6 weeks were proposed. The exercise intensity of exercise corresponds to target heart rate at ventilatory threshold measured during incremental exercise test. Training at this intensity allowed us to individualize effort for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary mild to severe COPD patients

Exclusion Criteria:

* Neuromuscular disease
* Chronic heart failure
* Renal diseases
* Liver diseases
* Obesity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cellular effects of exercise training at the ventilatory threshold intensity | 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maurice MH Hayot, MCU-PH, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- France (2):
  - Clinique du Souffle La Vallonie, Lodève
  - Clinique du Souffle la Solane, Osséja